CLINICAL TRIAL: NCT03635177
Title: Effect of Remote Ischemic Conditioning on Vascular Health in Stroke Patients
Acronym: VISP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Ylva Hellsten, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RIC stroke
Record Dates: First submitted 2018-07-26; First posted 2018-08-17 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Stroke, Lacunar
MeSH Terms: conditions — Stroke, Lacunar

STUDY DESIGN:
Intervention Model Description: The patients will undergo two weeks of the intervention and two weeks of controlperiod, separated by three weeks. The intervention consists of inflating a cuff on the upperarm to 200 mmHg for 4 x 5 minutes, performed every day. The control period includes no specific intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote ischemic conditioning (Experimental): The participant will conduct remote ischemic preconditioning by use of an automated cuff device placed on the upper arm which inflates to 200 mmHg and occludes blood flow. The procedure is conducted on one arm 4 x 5 min per day. Each 5 min occlusion period is interspersed by 5 min.
  Interventions: Procedure: Remote ischemic conditioning
- Sham occlusion (Sham Comparator): The participant will conduct a sham procedure of remote ischemic preconditioning by use of an automated cuff device placed on the upper arm which inflates minimally and does not occlude blood flow. The procedure is conducted on one arm 4 x 5 min per day. Each 5 min of sham occlusion is interspersed by 5 min.
  Interventions: Procedure: Remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Four weeks of daily ischemic conditioning and four weeks of sham ischemic conditioning in a cross over design
  Other Names: Sham remote ischemic conditioning

SUMMARY:
The main aim of the current study is to assess cardiovascular effects of remote ischemic conditioning in patients who have suffered from stroke. A group of stroke patients will be subjected to four weeks of daily remote ischemic conditioning and four weeks of placebo and vascular function is assessed as a primary outcome.

DETAILED DESCRIPTION:
Remote ischemic preconditioning (RIC) has been shown to reduce myocardial damage in association with a myocardial infarct but less is known about the potential effects on vascular function in patients who have suffered a stroke. RIC is a procedure by which blood flow to a limb is repeatedly occluded during a short period by an inflatable cuff. This project evaluates the effect of a two week period with RIC on vascular function and cerebral blood flow velocity as well as on factors associated with blood clot formation in patients who have suffered a stroke. The study also aims to provide mechanistic insight into the beneficial effects of the RIC procedure.

Subjects are patients who within the past five years have suffered from lacunar infarct. The study is of a cross-over design with two weeks of homebased RIC treatment and two weeks of control period in a randomized order. Before and after the experimental periods the subjects undergo a number of tests assessing general health status, vascular function and cerebral blood flow velocity. Skeletal muscle samples are obtained for the determination of selected proteins related to vascular function and angiogenesis and blood samples are obtained for the determination of platelet function.

.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms and corresponding computer tomographytomography/magnetic resonance (CT/MR)-scanning results for lacunar infarct within past five years.
* Small vessel disease stroke (lacunar infarct) is defined by the TOAST criteria

Exclusion Criteria:

Clinical significant carotid stenosis. Cardioembolic stroke

* Clinically significant chronic diseases other than lacunar infarct and associated factors
* Current or past smoker within the past ten years
* Current treatment with beta-blockers, peroral steroids or NSAIDS
* Alcohol- or drug-addiction.
* Pregnant or lactating.
* Inability to understand the content of the study information provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilation | Change from baseline to 4 weeks
  Assessment of brachial artery dilation after 5 min occlusion of upper arm by cuff

SECONDARY OUTCOMES:
Cerebral vascular function-visual task | Change from baseline to 4 weeks
  Assessment of change in cerebral blood flow velocity with visual task
Cerebral vascular function- motorparadigm task | Change from baseline to 4 weeks
  Assessment of change in cerebral blood flow velocity with motorparadigm task
Skeletal muscle blood flow | Change from baseline to 4 weeks
  Femoral arterial blood flow measured at rest and during one leg knee extensor exercise
Platelet reactivity | Change from baseline to 4 weeks
  Platelet reactivity is assessed in platelets isolated from blood samples
Blood clot structure-gel point | Change from baseline to 4 weeks
  Blood clot structure is assessed by gel point
Blood clot structure-fractal analysis | Change from baseline to 4 weeks
  Blood clot structure is assessed by fractal analysis
Skeletal muscle proteins | Change from baseline to 4 weeks
  Proteins associated with angiogenesis and vascular function are assessed in skeletal muscle samples obtained from the thigh muscle
Plasma proteins | Change from baseline to 4 weeks
  Protein amount is determined in plasma
Plasma lipids | Change from baseline to 4 weeks
  Lipid concentration is determined in plasma
Oral glucose tolerance test (OGTT) | Change from baseline to 4 weeks
  An oral glucose tolerance test is conducted by assesment of blood glucose and insulin before and after ingestion of glucose
Body composition | Change from baseline to 4 weeks
  Body composition is assessed by dual energy x-ray absorptiometry

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - University of Copenhagen, Copenhagen
  - Department of Neurology, Herlev Hospital, Herlev

REFERENCES:
- [Derived] Norregaard LB, Wickham KA, Jeppesen JS, Rytter N, Christoffersen LC, Gliemann L, Lawrence M, Evans PA, Kruuse C, Hellsten Y. Exercise transiently increases the density of incipient blood clots in antiplatelet-treated lacunar stroke patients. Thromb J. 2024 Apr 5;22(1):35. doi: 10.1186/s12959-024-00604-9. PMID 38581046